CLINICAL TRIAL: NCT01433653
Title: Randomized Controlled Clinical Trial of Cognitive Behavioral Therapy for Complicated Grief
Brief Title: Cognitive Behavioral Therapy for Complicated Grief
Acronym: CG-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Rita Rosner, Prof. Dr. Rita Rosner, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: LMU-KlinPsy001
Record Dates: First submitted 2011-07-18; First posted 2011-09-14 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Grief
Keywords: Comorbid; Complicated
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CG-CBT (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Complicated Grief
- wait list control (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Complicated Grief — Manualized CBT with 25 sessions, once a week. Key elements are exposition and cognitive restructuring.
  Arms: CG-CBT

SUMMARY:
The purpose of this study is to determine whether cognitive behavioral therapy (CG-CBT) for complicated grief is superior to wait list condition in patients with comorbid complicated grief. To evaluate the effect pre-post changes for patients in the CG-CBT-group will be compared to changes in the wait list group.

ELIGIBILITY:
Inclusion Criteria:

* age complicated grief diagnosis

Exclusion Criteria:

* acute suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
PG-13 (Prolonged Grief Interview - 13 Item version) | Change between intake (t1) and end of treatment (t2) in complicated grief severity within 5 months. t1= before treatment or wait list begins, t2 = 4 months after t1 (end of treatment, end of waitlist), t3 = follow-up (1.5 years after t2)

SECONDARY OUTCOMES:
Symptom Checklist 90 revised (SCL-90R; Subscale General Symptom Index, GSI) | Change between intake (t1) and end of treatment (t2) in general distress symptoms within 5 months. t1= before treatment or wait list begins, t2 = 4 months after t1 (end of treatment, end of waitlist), t3 = follow-up (1.5 years after t2)
Comorbid Diagnoses by DIA-X-Interview | Change between intake (t1) and end of treatment (t2) in number of comorbid psychiatric diagnoses within 5 months; t1= before treatment or wait list begins, t2 = 4 months after t1 (end of treatment, end of waitlist), t3 = follow-up (1.5 years after t2)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Rosner, Dr. phil., Principal Investigator — LMU
Locations (1):
- LMU, Munich, Germany

REFERENCES:
- [Result] Rosner R, Pfoh G, Kotoucova M, Hagl M. Efficacy of an outpatient treatment for prolonged grief disorder: a randomized controlled clinical trial. J Affect Disord. 2014;167:56-63. doi: 10.1016/j.jad.2014.05.035. Epub 2014 Jun 2. PMID 25082115
- [Result] Rosner R, Bartl H, Pfoh G, Kotoucova M, Hagl M. Efficacy of an integrative CBT for prolonged grief disorder: A long-term follow-up. J Affect Disord. 2015 Sep 1;183:106-12. doi: 10.1016/j.jad.2015.04.051. Epub 2015 May 8. PMID 26001670